CLINICAL TRIAL: NCT02003040
Title: Role of the Mespere Venus 1000 in Predicting Heart Failure Hospital Readmissions
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Mespere Lifesciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: STP-9000011
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: ADHF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- St. Michael's Hospital Patients: Patients admitted to the Cardiology ward at St Michael's Hospital with a main diagnosis of acute decompensated heart failure
  Interventions: Device: Mespere Venus 1000 CVP System

INTERVENTIONS:
Device: Mespere Venus 1000 CVP System — An adhesive patch (connected to the Mespere Venus 1000 System) is placed on the neck of the subject. A CVP measurement is recorded at time of patient's hospital admission and discharge. CVP readings will remain concealed from the treating team.

SUMMARY:
The purpose of this study is to investigate the utility of Venus 1000 in predicting 30-day hospital readmissions for acute decompensated heart failure. Secondary outcomes will include correlation with NT-proBNP and weight both at admission and discharge from hospital

DETAILED DESCRIPTION:
Rehospitalizations for heart failure have been linked to poor clinical outcomes, rates remain high despite different attempts to decrease them . Clinical indicators of volume congestion at time of discharge are associated with increased rates of readmission . Clinical evaluation of volume status remains the gold standard in determination of readiness and timing of hospital discharge, however identification of persistent congestion might prove difficult .

Assessment of the right atrial pressure can be done non-invasively at the bedside; however, precision and accuracy of this method are variable . Echocardiography is a valuable tool in the estimation of elevated central pressure , this, however is time consuming and requires trained personnel. While invasive measurements provide accurate estimation of central venous pressure, it is an impractical approach in most patients, notwithstanding the risks associated with the insertion of a catheter into the central circulation .

Since a significant proportion of readmitted patients return to hospital with congestive symptoms, attempts have been made to improve our ability to assess volume status . Current clinical evidence suggests that BNP-guided management of patients with congestive heart failure can decrease all-cause mortality and heart failure rehospitalization. However, biological variation for natriuretic peptides is high , and optimal targets are difficult to determine in individual patients.

The Mespere Venus 1000 system is a non-invasive tool that has previously shown reliable correlation and accuracy with central venous pressure obtained invasively in the catheterization laboratory and good correlation with jugular venous pressure at the bedside.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Patient admitted to St. Michael's Hospital with a main clinical diagnosis of decompensated heart failure.
* Signed informed consent

Exclusion Criteria:

* Lack of patient consent.
* Presence of known AV dialysis fistula.
* Allergy to adhesive tape from Mespere Venus 1000 system.
* Known central vein stenosis.
* Ongoing photodynamic therapy.
* Assisted ventilation.
* Associated acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Cardiology ward at St Michael's Hospital with a main diagnosis of acute decompensated heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in non-invasive central venous pressure (NICVP) at time of hospital discharge | time of hospital admission (baseline) and time of hospital discharge
  To determine if NICVP (taken at time of hospital admission and discharge) from the Mespere Venus 1000 CVP System can predict 30-day hospital readmissions for acute decompensated heart failure.

SECONDARY OUTCOMES:
NT-proBNP | 1 visit
  To investigate if there's a correlation between CVP measurements from the Mespere Venus 1000 CVP System and NT-proBNP at time of hospital admission and discharge
Patient's weight | 1 visit
  To investigate if there's a correlation between CVP measurements from the Mespere Venus 1000 CVP System and weight change at time of hospital admission and discharge

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Al-Hesayen, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada